CLINICAL TRIAL: NCT00979524
Title: Addressing Mental Health in African American Job Training Adolescents and Young Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: U48DP001919-01 (NIH)
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Depression
Keywords: Depressive symptoms; Mental health services; Adolescents; Young adults; African-American
MeSH Terms: conditions — Depression | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive Mental Health Services (Experimental): Intervention group participants will receive an array of mental health education and services based on their level of need. Study participants will fall into low, moderate, or elevated risk based on results of baseline screening. Services will be provided to each group as specified below. Low risk group: (a) Initial meeting with one of the licensed clinical social workers (LCSW-C), (b) education activities to promote knowledge and change attitudes around mental health; Moderate risk group: (a) Initial meeting with one of the licensed clinical social workers (LCSW-C), (b) Short-term mental health services delivered by the LCSW-C, (c) Depression prevention intervention, (d) Education activities to promote knowledge and change attitudes around mental health; High risk group: (a) Initial meeting with one of the licensed clinical social workers (LCSW-C), (b) Mental health treatment services, (c) Education activities to promote knowledge and change attitudes around mental health.
  Interventions: Behavioral: Comprehensive Mental Health Services and Supports
- Usual Care (Employment Training Services) (Active Comparator): Newly enrolling Westside YO members will receive "usual care" services, which constitute a moderate level of mental health services and supports. The usual care services related to mental health at the Westside will include (1) the ACASI screen for all newly enrolling Westside YO members, (2) the initial visit with a LCSW-C, and (3) mental health training for Westside Case Advocates. More extensive mental health educational activities and services (e.g., additional sessions with LCSW-C, SOS Club) provided to the intervention group will not be available at the Westside YO Center during the initial study period. Also, Eastside Case Advocates will receive more extensive and ongoing mental health training.
  Interventions: Behavioral: Comprehensive Mental Health Services and Supports

INTERVENTIONS:
Behavioral: Comprehensive Mental Health Services and Supports — This study uses a quasi-experimental design to test the efficacy of a comprehensive mental health intervention to improve the mental health and employment outcomes of young adults (18-24) enrolling in the Eastside YO Program. Newly enrolling Eastside YO members will receive an array of mental health education and services based on level of need and serve as this study's intervention group. Newly enrolling Westside YO members will receive "usual care" services delivered by the staff at the Westside YO Program and serve as this study's comparison group.

SUMMARY:
This project's focus is twofold-to change the culture of an employment training program for adolescents and young adults (Youth Opportunities, or "YO") to more fully address the many mental health issues faced by its participants and to expand and improve the quantity and quality of mental health services for YO members. Four project components have been carefully selected to address the mental health issues of YO members: (1) Mental health education/training for YO staff and peer leaders, (2) Mental health education activities for YO members, (3) mental health screening on all newly enrolling YO members, and (4) comprehensive mental health services for YO members. These project components will be implemented at the HEBCAC YO Program (subsequently referred to as "Eastside" YO), with the Westside YO Program initially participating as a control site. Researchers at the Johns Hopkins University Center for Adolescent Health, led by Dr. Darius Tandon of the Department of Pediatrics, will conduct the research examining the effectiveness of these mental health services and supports.

There are four project objectives. First, the proposed activities will increase YO members' knowledge of mental health resources and decrease stigma associated with seeking mental health services. Second, the investigators will see an increase in YO members' receipt of needed mental health services. Third, the investigators will see improvement in YO members' mental health. Fourth, as a result of their improved mental health, YO members will more actively engage in YO program activities and achieve more key program milestones (e.g., GED completion). These objectives are sequential, with later objectives predicated on the achievement of earlier ones.

ELIGIBILITY:
Inclusion Criteria:

* All newly enrolling Eastside and Westside YO members during the study period will be eligible for study participation.

Exclusion Criteria:

* We will not enroll YO members currently in foster care in this study.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 782 (Actual)
Dates: Start 2008-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | November 2008-November 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore City Eastside and Westside Youth Opportunity Centers, Baltimore, Maryland, United States